CLINICAL TRIAL: NCT06373809
Title: Diabetic Foot: Treatment of Chronic Ulcers and Neuropathy With Transplantation of Placenta Derived Stem Cells (PDSC) - A Dose Escalation Safety and Exploratory Efficacy Study
Brief Title: Placenta Derived Stem Cells for Treating of Chronic Ulcers and Neuropathy
Acronym: PDSC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Michael H Carstens (Other)
Collaborators: Ministerio de Salud de Nicaragua (Unknown); Wake Forest Institute for Regenerative Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDSC1970222
Record Dates: First submitted 2024-04-08; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Diabetic Foot; Diabetic Neuropathies; Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot; Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: Prospective an open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot Ulcer (Experimental): The intervention at the foot in group 1 will be carried out by PDSC suspension in 60cc Lactated Ringer's (LR) solution. There will be 3 sequential blocks of subjects with increasing PDSC dose:
  * Block 1 (4 subjects) Total dosage (30 x 10*6 cells)
  * Block 2 (3 subjects) Total dosage (40 x 10*6 cells)
  * Block 3 (3 subjects) Total dosage (60 x 10*6 cells)
  Administration to the ipsilateral foot / ankle in group 1 is performed by four injection sites: (1) 20 cc into the wound bed, (2) 20 cc subcutaneously around the perimeter of the wound, (3) 10 cc along the tibialis posterior pathway at the ankle prior to entry into the plantar surface, and (4) 10 cc along the tibialis anterior / dorsal foot pathway from the ankle to the dorsum of the foot.
  Interventions: Biological: Transplantation of Placenta Derived Stem Cells
- Foot Ulcer and Leg neurophathy (Experimental): Dosing to the leg in group 2 will be carried out by PDSC suspension of the dose in 90cc LR solution, which will be divided equally among the three compartments of the leg. There will be 3 sequential blocks of subjects with increasing PDSC dose:
  * Block 1 (4 subjects) Total dosage (30 x 10*6 cells)
  * Block 2 (3 subjects) Total dosage (40 x 10*6 cells)
  * Block 3 (3 subjects) Total dosage (60 x 10*6 cells)
  Administration to the leg will be performed through a 5 mm incision in each compartment (anterior, posterior, and lateral) at a level lower than the anterior tibial tubercle plane. These incisions will allow the introduction of a liposuction cannula of 3-4 mm in diameter and 20 cc in length, with an aroma tip and a single port that will be passed distally until the limit of the compartment is reached and, from there, the PDSCs will be injected retrograde throughout the compartment.
  Interventions: Biological: Transplantation of Placenta Derived Stem Cells

INTERVENTIONS:
Biological: Transplantation of Placenta Derived Stem Cells — Subcutaneously administered placental-derived SVF / PDSC cells in foot, ankle, and calf tissues in 20 DFU patients

SUMMARY:
This is an initial dose escalation safety and exploratory efficacy study to treat two groups of subjects with critically sized diabetic wounds and diabetic neuropathy using placental-derived stem cells (PDSC) transplanted by injection into soft tissues of the lower limb. Its primary objective is safety assessment and its secondary objective is determining optimum PDSC safe dose. Group 1 will receive implantation of cells in the ulcer, in the ulcer bed, and along the distal arterial vessels that supply blood to the foot. Group 2 will follow the same protocol for the foot but will have an additional dose of cells implanted in the anterior and posterior compartments of the same leg to determine the impact on peripheral neuropathy. Dose escalation and safety will be documented. Exploratory measures of efficacy include: ulcer healing, hemodynamic and anatomical effects on the arteries of the foot, and changes in the sensory perceptions of the foot.

DETAILED DESCRIPTION:
Diabetes mellitus is a global public health threat, with a projected global cost of US $825 billion by 2030 and $845 billion by 2045 (International Diabetes Federation). Angiopathy (macrovascular and / or microvascular) and neuropathy secondary to disease sets the stage for diabetic foot ulceration (DFU) by initiating cycles of inflammation, ulceration, infection, and hospitalization, often resulting in amputation. DFU in the context of a combined neuro-ischemic disease has a worse outcome. In the United States, 54% of all amputations are related to diabetes, and in 85% of cases, the trigger is a DFU, costing $9 to $13 billion per year.

Peripheral vascular disease (PVD) due to arteriosclerosis is also a known cause of ischemic ulcers and is also an aggravating condition of DFU. PVD, either alone or in combination with diabetes, often culminates in amputations and recurrent ulcers that do not heal. Approximately 50% of patients with DFU have concurrent vascular disease. As surgical revascularization is not always feasible in these patients, there is an urgent need to develop alternative therapies capable of improving the blood supply to the ischemic foot.

Cell-based therapies have gained attention as viable options to provide the elements necessary to help restore damaged vessels while inducing the formation of new ones. Cell products may contain endothelial progenitor cells (EPC) and / or mesenchymal stem / stromal cells (MSC), both critical during vascular repair and formation given the structural involvement of EPC and the documented pro-angiogenic activity of MSC. Based on the capabilities of the documented individual cell types for EPC and MSC, the use of a combinatorial cell approach in the same product constitutes an interesting alternative for treating vascular disease. Multiple small clinical studies have used autologous or allogeneic bone marrow mononuclear cells (MNC), either directly after bone marrow extraction or after tissue culture, to treat critical limb ischemia. In general, the therapy resulted in an improvement in symptoms, such as a decrease in pain, and in some studies the ankle / arm index and / or tissue oxygenation improved.

Adipose-derived vascular stromal fraction (AD-SVF) is a viable option to treat vascular disease, given its enrichment in EPC and higher MSC titers compared to other sources, e.g., bone marrow. Logistical advantages complement this key multi-phenotypic display as SVF cells can be obtained from same-day processing of easily accessible harvested adipose tissue without the need for a Good Manufacturing Practice (GMP) processing facility to manufacture an MSC-based product, thus making SVF a "point of care" therapy.

It is difficult to treat vascular disease and chronic ulcers caused by PVD and / or diabetes in resource-poor countries like Nicaragua. Most patients are unable to maintain a limited weight bearing or non-ambulatory state due to the economic imperative of working. Patients often have to travel long distances on poor road conditions to obtain medical care. Revascularization procedures are not economically possible for the majority of the Nicaraguan population. Additionally, advanced stem cell procedures that require cell processing facilities pose significant logistical and economic challenges.

In such conditions, non-healing ischemic wounds present patients and clinicians with undesirable options: chronic pain and risk of infection or amputation. Given these factors, the Nicaraguan Ministry of Health authorized a pilot study in 2014 to evaluate the potential value of freshly isolated autologous adipose-derived SVF cells as an alternative and cost-effective form of treatment for PVD caused by arteriosclerosis and / or diabetes.

Studies with AD-SVF for vascular insufficiency in Nicaragua

Given the clinical challenge of peripheral vascular disease in Nicaragua, the Ministry of Health and Assistance (MINSA) approved two successive clinical studies to evaluate the safety, efficacy, and applicability of AD-SVF cells for this indication. Both studies were open-label and non-randomized, and SVF cells were injected into affected tissues. The studies were carried out in the teaching hospitals of the MINSA in León (Hospital Escuela Oscar Danilo Rosales Argüello, HEODRA), in Managua (Hospital Escuela Manolo Morales, HEMM) and in Matagalpa (Hospital Escuela Cesar Amador Molina, HECAM).

Clinical study 1a (initial phase): Non-reconstructable peripheral vascular disease of the lower extremity in ten patients treated with adipose-derived stromal vascular fraction cells.

Clinical study 1b (follow-up phase): Adipose-derived stromal vascular fraction (SVF) cells for the treatment of non-rebuildable peripheral vascular disease in patients with critical limb ischemia: a 6-year follow-up showing long-lasting results.

Clinical study 2: Treatment of chronic diabetic foot ulcers with injections of stromal vascular fraction cells derived from adipose tissue: safety and evidence of efficacy at one year.

The key lessons learned from the previous studies are as follows:

* Local administration of SVF cells produces accelerated wound healing.
* SVF cells are capable of improving arterial blood flow under otherwise ischemic conditions.
* The administration of SVF along the path of the distal arteries supplying the foot (tibialis anterior and tibialis posterior) is associated with changes in the waveform and flow velocity compatible with the induction of new vessels and the reduction of distal resistance.

Objectives of the study

Primary Objective: To determine the safety of transplantation of PDSCs in the lower limb in 20 patients with diabetes and critical size ulcers (≥10cm2)

Exploratory Objective- To determine if PDSC improve diabetes-associated lower extremity pathophysiology

* Document wound healing
* Quantify flow parameters and elasticity of pedal arteries.
* Document sensation in the diabetic foot

Study hypotheses

Primary hypothesis - Transplantation of PDSCs in the diabetic foot is safe

Exploratory Hypothesis - PDSC improve diabetes-associated lower extremity pathophysiology

Subcutaneously administered placental-derived SVF / PDSC cells in foot, ankle, and calf tissues (as indicated) in 20 DFU patients are effective as follows:

* PDSCs, by increasing the distal vessels of the foot, can increase the flow rates measured in the tibialis anterior, dorsalis of the foot, and tibialis posterior.
* PDSCs when applied near the arteries of the foot affected by diabetes can exert a trophic effect on fibrotic arterial walls.
* PDSCs, by exerting local anti-inflammatory and neo-angiogenesis effects, can improve the sensory function of the nerves that serve the foot: fibula, sural and posterior tibialis.

To assess the possible effects on neurological sensation of PDSCs administered subcutaneously in the tissues of the foot, ankle, and calf (as indicated) in 10 patients with DFU

* PDSCs, due to their angiogenic effect, can improve / increase microcirculation to the peripheral nerves that serve the foot and consequently improve their function.
* PDSCs, due to their antifibrotic effect, can reduce perineural fibrosis and consequently improve its function.

Study design

Format

* Prospective
* Open label
* Primary Endpoint: safety and dose at 3 months, 6 months, 9 months, 1 year
* Secondary Endpoint: improvements in diabetes associated pathophysiology at 3 months, 6 months, 9 months, 1 year
* Intervention: PDSC administration to two subject groups - application of PDSCs to the foot with and without to the compartments of the leg
* Masking: open label
* Main objective: Safety
* Exploratory objective: improvement in diabetes associated pathophysiology
* Dosage: dose escalation

Diagnosis and selection of patients

It is proposed to study 20 patients with a diagnosis of peripheral vascular insufficiency due to diabetes mellitus, which manifests as an ulcer (for more than 2 months) and with vascular anatomy to the point that they are not candidates for surgical intervention.

The number of patients in the two groups is based upon a standard approach to dose escalation. The study should provide insights into efficacy to be used in subsequent clinical trials but is not powered for an efficacy trial.

Study procedures

Processing, delivery and storage of PDSC

PDSC will be prepared from the cell bank in Wake Forest Institute for Regenerative Medicine (WFIRM) as indicated above. The technical aspects of the preparation and the associated costs are detailed in Annex 1. Transportation to Nicaragua will be carried out by World Carrier with direct delivery to the National Center for Diagnosis and Reference [Centro Nacional de Diagnostico y Referencia (CNDR)] at the Concepción Palacios National Health Complex in Managua.

PDSCs will be transported from the -80 ° freezer in CNDR. The freezer is temperature monitored and linked to an active alarm system. PDSCs will be transported from the -80 ° freezer in CNDR to the treatment site on the day of the intervention. PDSC will be used within 2 hours of warming. Cells not used in a timely fashion will be destroyed and their destruction will be recorded as will the reason that they were not used.

Study Structure

Potential subjects will be identified from the León and Matagalpa regions, then will be evaluated by the surgical services of the following hospitals: (1) Hospital Escuela Oscar Danilo Rosales Arguello, León (HEODRA); (2) Hospital Escuela Cesar Amador Molina, Matagalpa (HECAM).

ELIGIBILITY:
Inclusion Criteria:

* well-controlled diabetes
* unilateral wound that exceeds an area ≥ 10 cm2, present for > 3 months
* not candidates for surgical reconstruction
* able to understand and provide informed consent
* an additional diagnosis of peripheral arteriosclerosis is allowed.

Exclusion Criteria:

* presence of a disease that prohibits surgical intervention
* inadequate medical control of diabetes
* smoking, substance abuse within 3 months of the onset of the study
* inability to understand or fulfill the objectives and responsibilities of the study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Foot Ulcer Healing | Baseline, 3, 6, 9 and 12 months post treatment.
  Percent closure based on changes in ulcer size dimensions in square cm.

SECONDARY OUTCOMES:
Fine Touch Sensation: Documenting diabetes-associated lower extremity pathophysiology changes. | Baseline, 3, 6, 9 and 12 months post treatment.
  Semmes-Weinstein scores to document sensation threshold
Vibration: Documenting diabetes-associated lower extremity pathophysiology changes. | Baseline, 3, 6, 9 and 12 months post treatment.
  Horwell neurothesiometer scores to document vibration threshold

CONTACTS AND LOCATIONS:
Locations (2):
- Nicaragua (2):
  - Hospital Escuela Oscar Danilo Rosales Arguello (HEODRA), León, León Department
  - Hospital Escuela Cesar Amador Molina, Matagalpa

REFERENCES:
- [Background] Amos PJ, Shang H, Bailey AM, Taylor A, Katz AJ, Peirce SM. IFATS collection: The role of human adipose-derived stromal cells in inflammatory microvascular remodeling and evidence of a perivascular phenotype. Stem Cells. 2008 Oct;26(10):2682-90. doi: 10.1634/stemcells.2008-0030. Epub 2008 Apr 24. PMID 18436860
- [Background] Armulik A, Genove G, Betsholtz C. Pericytes: developmental, physiological, and pathological perspectives, problems, and promises. Dev Cell. 2011 Aug 16;21(2):193-215. doi: 10.1016/j.devcel.2011.07.001. PMID 21839917
- [Background] Arnberg F, Lundberg J, Olsson A, Samen E, Jaff N, Jussing E, Dahlen U, Nava S, Axelsson R, Ringden O, Kaipe H, Holmin S. Intra-arterial Administration of Placenta-Derived Decidual Stromal Cells to the Superior Mesenteric Artery in the Rabbit: Distribution of Cells, Feasibility, and Safety. Cell Transplant. 2016;25(2):401-10. doi: 10.3727/096368915X688191. Epub 2015 May 13. PMID 25976072
- [Background] Bainbridge DR, Ellis SA, Sargent IL. HLA-G suppresses proliferation of CD4(+) T-lymphocytes. J Reprod Immunol. 2000 Aug;48(1):17-26. doi: 10.1016/s0165-0378(00)00070-x. PMID 10996380
- [Background] Berishvili E, Kaiser L, Cohen M, Berney T, Scholz H, Floisand Y, Mattsson J. Treatment of COVID-19 Pneumonia: the Case for Placenta-derived Cell Therapy. Stem Cell Rev Rep. 2021 Feb;17(1):63-70. doi: 10.1007/s12015-020-10004-x. PMID 32696426
- [Background] Bishop PD, Feiten LE, Ouriel K, Nassoiy SP, Pavkov ML, Clair DG, Kashyap VS. Arterial calcification increases in distal arteries in patients with peripheral arterial disease. Ann Vasc Surg. 2008 Nov;22(6):799-805. doi: 10.1016/j.avsg.2008.04.008. Epub 2008 Jul 21. PMID 18640812
- [Background] Bourin P, Bunnell BA, Casteilla L, Dominici M, Katz AJ, March KL, Redl H, Rubin JP, Yoshimura K, Gimble JM. Stromal cells from the adipose tissue-derived stromal vascular fraction and culture expanded adipose tissue-derived stromal/stem cells: a joint statement of the International Federation for Adipose Therapeutics and Science (IFATS) and the International Society for Cellular Therapy (ISCT). Cytotherapy. 2013 Jun;15(6):641-8. doi: 10.1016/j.jcyt.2013.02.006. Epub 2013 Apr 6. PMID 23570660
- [Background] Bura A, Planat-Benard V, Bourin P, Silvestre JS, Gross F, Grolleau JL, Saint-Lebese B, Peyrafitte JA, Fleury S, Gadelorge M, Taurand M, Dupuis-Coronas S, Leobon B, Casteilla L. Phase I trial: the use of autologous cultured adipose-derived stroma/stem cells to treat patients with non-revascularizable critical limb ischemia. Cytotherapy. 2014 Feb;16(2):245-57. doi: 10.1016/j.jcyt.2013.11.011. PMID 24438903
- [Background] Caplan AI, Correa D. The MSC: an injury drugstore. Cell Stem Cell. 2011 Jul 8;9(1):11-5. doi: 10.1016/j.stem.2011.06.008. PMID 21726829
- [Background] Carstens MH, Correa D, Llull R, Gomez A, Turner E, Valladares S. Subcutanous reconstruction of hand dorsum for late sequelae of burn scars using stromal vascular fractions (SVF). CellR4 2015; 3; e1675.
- [Background] Carstens MH, Gomez A, Cortes R, Turner E, Perez C, Ocon M, Correa D. Non-reconstructable peripheral vascular disease of the lower extremity in ten patients treated with adipose-derived stromal vascular fraction cells. Stem Cell Res. 2017 Jan;18:14-21. doi: 10.1016/j.scr.2016.12.001. Epub 2016 Dec 8. PMID 27984756
- [Background] Carstens MH, Mendieta M, Perez C, Villareal E, Garcia R. Assisted Salvage of Ischemic Fasciocutaneous Flap Using Adipose-Derived Mesenchymal Stem Cells: In-Situ Revascularization. Aesthet Surg J. 2017 Jul 1;37(suppl_3):S38-S45. doi: 10.1093/asj/sjx052. PMID 29025216
- [Background] Carstens MH, Pérez M, Briceño H, Valladares S, Correa D. Treatment of late sequelae of burn scar fibrosis with adipose-derived stromal vascular fraction (SVF) cells: a case series. CellR4 2017; 5: e2404.